CLINICAL TRIAL: NCT05296811
Title: Lateral Arm Free Flap for Reconstruction of the Oral Cavity and Head and Neck Soft Tissue Defects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hassan harby mohamed (Other)
Responsible Party: Sponsor-Investigator, hassan harby mohamed, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Lateral Arm Free Flap
Record Dates: First submitted 2022-03-06; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lateral Arm Free Flap — Primary Reconstruction of intraoral defects by use of Lateral Arm Free Flap.

SUMMARY:
The excision of oral cancers causes extensive impairment of the oral cavity soft tissue. Complete excision of the tumors is vital, and the reconstruction of the resected area influences not only the postoperative recovery period of patients but also physiological functions such as swallowing, phonation function ,daily activities and psychosocial impact.

Oral and maxillofacial surgeons are faced with the task of reconstructing the affected area to reduce these problems as much as possible.

In 1982, Song introduced the lateral arm flap (LAF). Since this time, its used in surgical repairs of oral defects, But the specific subject of publications generally restricted to a small number of cases.

LAF is a thin and pliable flap with consistent anatomy and a high success rate. It is also claimed that there is no risk of vascular compromise to the arm

DETAILED DESCRIPTION:
reconstruction of oral , head and neck defects with Lateral Arm Free Flap

ELIGIBILITY:
Inclusion Criteria:

1. All patients post glossectomy.
2. Patients post maxillectomy with malignant maxillary swelling with no distant metastases.
3. All patients which defect after surgery for head and neck neoplasia.

Exclusion Criteria:

* 1. Small defect post excision can be closed directly 2. medically unfit patients

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of recurrence | 3 month
  reconstruction of defects in head and neck post surgical excision by lateral arm free flap and early detection of recurrence by CT neck.

CONTACTS AND LOCATIONS:
Overall Officials: hassan harby, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Nahabedian MY, Deune EG, Manson PN. Utility of the lateral arm flap in head and neck reconstruction. Ann Plast Surg. 2001 May;46(5):501-5. doi: 10.1097/00000637-200105000-00008. PMID 11352423